CLINICAL TRIAL: NCT01967953
Title: Ex-Vivo Lung Perfusion to Improve Donor Lung Function and Increase the Number of Organs Available for Transplantation
Brief Title: Ex-Vivo Lung Perfusion to Increase the Number of Organs for Transplantation
Acronym: EVLP_MI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Franco Valenza, MD, Assistant Professor Anaesthesia and Intensive Care, Department of Pathophysiology and Transplantation, Università degli Studi di Milano, Policlinico Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EVLP_2011
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Disorder Related to Lung Transplantation; Brain Death; Graft Failure; Primary Graft Dysfunction
MeSH Terms: conditions — Brain Death; Primary Graft Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Group (No Intervention): Recipients of lungs procured from brain death donors deemed suitable for transplantation according to standard criteria.
  Events: lung procurement, cold storage on ice, transplantation.
- EVLP Group (Experimental): Recipients of marginal lungs procured from brain death donors and reconditioned with ex-vivo lung perfusion (EVLP).
  Events: lung procurement, cold storage on ice, reconditioning by EVLP, cold storage on ice, transplantation.
  Interventions: Procedure: EVLP Group

INTERVENTIONS:
Procedure: EVLP Group — EVLP technique: Steen solution; normothermia; low flow, open atrium, low hematocrit.
  Endpoints of EVLP assessment of lungs suitability: oxygenation, respiratory mechanics, pulmonary vascular resistance, chest X-ray, fibrobronchoscopy
  Arms: EVLP Group

SUMMARY:
The recent introduction of ex-vivo lung perfusion (EVLP) as a tool to evaluate and recondition lungs from marginal donors has opened a new era in the field of lung transplantation.

DETAILED DESCRIPTION:
Aim of the investigation: to compare the clinical outcome after transplantation of subjects receiving marginal lungs procured from brain death donors and reconditioned by EVLP, with that of subjects receiving lungs procured from standard donors.

ELIGIBILITY:
Inclusion criteria for donor lung:

1. Recipient to undergo single or bilateral Lung Transplantation
2. Donor arterial partial pressure of oxygen to fraction of inspired oxygen ratio (PaO2/FiO2) below 300 mmHg, or doubtful donor lung function

Exclusion criteria for donor lung:

1. Massive lung contusion
2. Aspiration
3. Pneumonia
4. Sepsis
5. Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Primary Graft Dysfunction 72 hours after lung transplantation (PGD72) | 72 hours
  Primary Graft Dysfunction 72 hours after transplantation (PGD72) definition: grade 3 according to the International Society of Heart and Lung Transplantation classification
30 day Mortality | 30 days

SECONDARY OUTCOMES:
Duration of mechanical ventilation after transplantation | 30 days
ICU length of stay after transplantation | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Franco Valenza, MD, Principal Investigator — Fondazione Ca' Granda IRCCS Ospedale Maggiore Policlinico Milan Italy
Locations (1):
- Fondazione Ca' Granda IRCCS Ospedale Maggiore Policlinico, Milan, Italy, Italy

REFERENCES:
- [Background] Cypel M, Yeung JC, Liu M, Anraku M, Chen F, Karolak W, Sato M, Laratta J, Azad S, Madonik M, Chow CW, Chaparro C, Hutcheon M, Singer LG, Slutsky AS, Yasufuku K, de Perrot M, Pierre AF, Waddell TK, Keshavjee S. Normothermic ex vivo lung perfusion in clinical lung transplantation. N Engl J Med. 2011 Apr 14;364(15):1431-40. doi: 10.1056/NEJMoa1014597. PMID 21488765
- [Background] Oto T, Levvey BJ, Whitford H, Griffiths AP, Kotsimbos T, Williams TJ, Snell GI. Feasibility and utility of a lung donor score: correlation with early post-transplant outcomes. Ann Thorac Surg. 2007 Jan;83(1):257-63. doi: 10.1016/j.athoracsur.2006.07.040. PMID 17184674
- [Background] Aigner C, Winkler G, Jaksch P, Seebacher G, Lang G, Taghavi S, Wisser W, Klepetko W. Extended donor criteria for lung transplantation--a clinical reality. Eur J Cardiothorac Surg. 2005 May;27(5):757-61. doi: 10.1016/j.ejcts.2005.01.024. PMID 15848310
- [Background] Steen S, Ingemansson R, Eriksson L, Pierre L, Algotsson L, Wierup P, Liao Q, Eyjolfsson A, Gustafsson R, Sjoberg T. First human transplantation of a nonacceptable donor lung after reconditioning ex vivo. Ann Thorac Surg. 2007 Jun;83(6):2191-4. doi: 10.1016/j.athoracsur.2007.01.033. PMID 17532422
- [Background] Valenza F, Rosso L, Coppola S, Froio S, Colombo J, Dossi R, Fumagalli J, Salice V, Pizzocri M, Conte G, Gatti S, Santambrogio L, Gattinoni L. beta-adrenergic agonist infusion during extracorporeal lung perfusion: effects on glucose concentration in the perfusion fluid and on lung function. J Heart Lung Transplant. 2012 May;31(5):524-30. doi: 10.1016/j.healun.2012.02.001. Epub 2012 Mar 3. PMID 22386450
- [Background] Botha P, Trivedi D, Weir CJ, Searl CP, Corris PA, Dark JH, Schueler SV. Extended donor criteria in lung transplantation: impact on organ allocation. J Thorac Cardiovasc Surg. 2006 May;131(5):1154-60. doi: 10.1016/j.jtcvs.2005.12.037. PMID 16678604
- [Background] Valenza F, Rosso L, Pizzocri M, Salice V, Umbrello M, Conte G, Stanzi A, Colombo J, Gatti S, Santambrogio L, Iapichino G, Gattinoni L. The consumption of glucose during ex vivo lung perfusion correlates with lung edema. Transplant Proc. 2011 May;43(4):993-6. doi: 10.1016/j.transproceed.2011.01.122. PMID 21620034
- [Derived] Valenza F, Rosso L, Coppola S, Froio S, Palleschi A, Tosi D, Mendogni P, Salice V, Ruggeri GM, Fumagalli J, Villa A, Nosotti M, Santambrogio L, Gattinoni L. Ex vivo lung perfusion to improve donor lung function and increase the number of organs available for transplantation. Transpl Int. 2014 Jun;27(6):553-61. doi: 10.1111/tri.12295. Epub 2014 Apr 4. PMID 24628890